CLINICAL TRIAL: NCT05426512
Title: Effect of Mechanical Loading on vBMD and Geometry in Patients With Primary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: EFSTATHIOS CHRONOPOULOS (Other)
Responsible Party: Sponsor-Investigator, EFSTATHIOS CHRONOPOULOS, Associate Professor in Orthopaedics at National and Kapodistrian University of Athens, Laboratory for Research of the Musculoskeletal System Director, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Other Study IDs: NKUAthens1
Record Dates: First submitted 2022-06-10; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Primary Hyperparthyroidism
- Postmenopausal women

SUMMARY:
In this study we aimed to evaluate the effect of primary hyperparathyroidism (PHPT) on bone geometry simultaneously at the tibia and the radius, peripheral bone sites with similar structure but subject to different loading conditions. This evaluation was made by comparing z-scores of bone parameters measured by peripheral quantitative computed tomography (pQCT).

DETAILED DESCRIPTION:
Postmenopausal women with primary hyperparathyroidism will be included in the study. The diagnosis of primary hyperparathyroidism is based on the high levels of parathyroid hormone and calcium.

Postmenopausal women with kidney failure, liver failure, malabsorption syndromes, women under medication that can affect the levels of the parathyroid hormone (lithium, thiazide diuretics) and calcium levels (oestrogen, loop diuretics, denosumab, bisphosphonates), corticosteroids, and women diagnosed with familial hypocalciuric hypercalcemia will be excluded from the study.

The control group has similar demographic characteristics and years of menopause with the patients that have primary hyperparathyroidism. Their calcium and parathyroid hormone levels are within the normal range and there is an absence of any secondary causes of osteoporosis.

The patients' medical files will be taken from the archives of the Laboratory for research of the Musculoskeletal System 'Th.Garofalidis', Medical School, National and Kapodistrian University of Athens, KAT General Hospital of Athens. The records of these patients will be used for the recording of the total calcium levels, parathyroid hormone levels, vitamin D, creatinine, albumin, alkaline phosphatase (ALP), along with bone mineral density at the lumbar spine and femur, with the use of dual-energy x-ray absorptiometry (DEXA). Moreover, pQCT measurements of bone parameters in the region 4% (trabecular bone) and 38% (cortical bone) at the tibia and in the region 4% (trabecular bone) and 20% (cortical bone) at the radius will be recorded. pQCT bone parameters that will be recorded include total bone mineral content (tot BMC), cortical bone mineral content (cort BMC), trabecular bone mineral content (trab BMC), total bone mineral density (tot BMD), cortical bone mineral density (cort BMD), trabecular bone mineral density (trab BMD), total area (tot AREA), trabecular area (trab AREA), cortical area (cort AREA), cortical thickness (cort THICK), endocortical and periosteal circumference (enco C and peri C) and calculation of SSI.

The primary endpoint of the study will be the comparison between the z-scores of the volumetric bone mineral density of the trabecular (trab BMD) and cortical bone (cort BMD) between the tibia and the radius. Secondary endpoints will be the differences between z-scores of the following variables in the region of the tibia and the radius. (trab BMC, cort BMC, trab AREA, cort AREA, cort THICK, endo C, peri C και SSI). Finally, the study will focus on if any differences between the z-scores are related to the severity of primary hyperparathyroidism, as it is defined by the levels of the parathyroid hormone and calcium.

ELIGIBILITY:
Inclusion Criteria:

Caucasian postmenopausal women with PHPT

Exclusion Criteria:

Chronic kidney disease (eGFR< 60 ml/min/1.73m2), Liver disease Malabsorption syndromes Rheumatic disease Women under medication that could affect aBMD or vBMD measurements, PTH, and /or calcium levels (lithium, thiazide/loop diuretics, estrogen, SERMS, denosumab, bisphosphonates) and corticosteroids

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Caucasian postmenopausal women with PHPT and healthy Caucasian postmenopausal women
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Effect of mechanical loading on vBMD and geometry in patients with primary hyperparathyroidism | Up to 24 weeks
  z-score for total volumetric bone mineral density (tot vBMD)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karlafti E, Dontas I, Lambrinoudaki I, Vlamis I, Lampropoulou-Adamidou K, Makris K, Trifonidi I, Galanos A, Trovas G, Chronopoulos E, Tournis S. Site specific differences in vBMD and geometry in postmenopausal women with primary hyperparathyroidism. Endocrine. 2024 Jan;83(1):205-213. doi: 10.1007/s12020-023-03491-8. Epub 2023 Aug 19. PMID 37597095